CLINICAL TRIAL: NCT03773744
Title: A Phase 1b, Multicenter, Open-label Trial of Oncolytic MG1 Expressing MAGE-A3 (MG1-MAGEA3) With Adenovirus Vaccine Expressing MAGE-A3 (Ad-MAGEA3), in Combination With Immune Modulating Therapy in Patients With Metastatic Melanoma or Previously Treated Cutaneous Squamous Cell Carcinoma
Brief Title: MG1-MAGEA3 With Ad-MAGEA3 and Pembrolizumab in Patients With Previously Treated Metastatic Melanoma or Cutaneous Squamous Cell Carcinoma
Acronym: Pelican
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: insufficient suitable drug supply
Sponsor: Turnstone Biologics, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ad/MG1-MAGEA3-003
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Melanoma; Squamous Cell Skin Carcinoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intravenous Dosing (Experimental): Low dose cyclophosphamide (300mg/ m2) at Day -3, then a fixed dose of Ad-MAGEA3 administered IM on study Day 1. Followed by one of 3 dose levels (escalation) of MG1-MAGEA3 administered as 2 intravenous (IV) doses at Day 15 and Day 18 and fixed dose pembrolizumab (200mg) beginning at either Week 6 or Day 1, depending on the cohort.
  Interventions: Drug: Ad-MAGEA3; Drug: MG1-MAGEA3; Drug: Pembrolizumab; Drug: Cyclophosphamide
- Arm 2: Intravenous followed by Intratumoral Dosing (Experimental): A fixed dose of Ad-MAGEA3 administered IM followed by Pembrolizumab on Day 1. MG1-MAGEA3 administered as an intravenous (IV) dose at Day 15, followed by intratumoral (IT) MG1-MAGEA3 on Day 22, Day 29, and Day 36. IT MG1-MAGEA3 booster injections may be continued every 3 weeks beginning at Day 43 (Week 6).
  Interventions: Drug: Ad-MAGEA3; Drug: MG1-MAGEA3; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Ad-MAGEA3 — Adenovirus vaccine expressing Melanoma-associated antigen 3 (MAGEA3), a tumor antigen
Drug: MG1-MAGEA3 — MG1 Maraba oncolytic virus expressing Melanoma-associated antigen 3 (MAGEA3), a tumor antigen
Drug: Pembrolizumab — monoclonal antibody; checkpoint inhibitor of PD1
  Other Names: Keytruda
Drug: Cyclophosphamide — low-dose chemotherapy
  Arms: Arm 1: Intravenous Dosing

SUMMARY:
This is a Phase 1b open-label dose escalation trial of Ad/MG1-MAGEA3 and Pembrolizumab in patients with Metastatic Melanoma or Cutaneous Squamous Cell Skin Cancer that has failed prior standard of care treatments. Upon determination of a Maximum Tolerated Dose (MTD) or Maximum Feasible Dose (MFD) the study will be expanded into up to 24 additional Metastatic Melanoma patients.

DETAILED DESCRIPTION:
This is a Phase 1b open-label dose escalation trial of Ad/MG1-MAGEA3 and Pembrolizumab in patients with Metastatic Melanoma or Cutaneous Squamous Cell Skin Cancer that has failed prior standard of care treatments. This study will consist of two arms where the dose will be increased independently until the maximum tolerated dose (MTD) / maximum feasible dose (MFD) is reached.

Arm 1 - Low-dose cyclophosphamide, followed by an Ad-MAGEA3 intramuscular (IM) prime, followed by intravenous (IV) administration of MG1-MAGEA3 and IV pembrolizumab.

Arm 2 - Ad-MAGEA3 IM injection as a prime, followed by IV administration of MG1-MAGEA3, followed by intratumoral (IT) injection of MG1-MAGEA3 into tumors and IV pembrolizumab.

In the Phase 1b Expansion for each arm, additional patients will be enrolled at the MTD/MDF as determined in Phase 1 in order to more thoroughly explore immune response, pharmacokinetics/dynamics, and safety for Malignant Melanoma patients who have failed standard therapies.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed diagnosis of locally advanced metastatic melanoma or cutaneous squamous cell carcinoma that has failed standard therapies
* For patients treated intratumorally, must have a lesion suitable for direct injection of MG1-MAGEA3
* Have at least one tumor amenable to biopsy
* Have measurable disease via RECIST 1.1 criteria
* Adequate organ function and performance status
* Additional inclusion criteria present

Exclusion Criteria:

* Prior treatment with any MAGE-A3 vaccine immunotherapy
* Prior systemic therapy for cancer within 4 weeks (8 weeks for lung radiation), and has recovered from chemo-related toxicities to Grade 1 or less
* Intolerant to prior PD1/PD-L1 therapy
* Requires use of anti-platelet or anti-coagulant therapy that cannot be safely suspended for per protocol biopsies or intra-tumoral injections.
* Known active CNS metastases and/or carcinomatous meningitis.
* Active autoimmune disease that has required systemic therapy in the past 2 years.
* Conditions likely to have resulted in splenic dysfunction.
* Known HIV/AIDS, active HBV or HCV infection.
* Additional Exclusion criteria exist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Ad/MG1-MAGEA3 administration in Melanoma or Squamous Cell Skin Carcinoma | 6 months
  Safety will be determined by assessing the severity and frequency of treatment emergent Adverse Events and clinical laboratory toxicity using NCI CTCAE v 5.0
Determine the maximum tolerated dose (MTD)/ maximum feasible dose (MFD) of Ad/MG1-MAGEA3 in Melanoma or Squamous Cell Skin Carcinoma | 5 weeks
  MTD/MFD of Ad/MG1-MAGEA3 administered by IV infusion alone and IV infusion followed by direct injection of tumor (IT injection) in Melanoma or Squamous Cell Skin Carcinoma

SECONDARY OUTCOMES:
Evaluate Overall Response | 2 years
  Determine the overall response rate (Partial Response (PR) + Complete Response (CR))
Evaluate Disease Control | 2 years
  Determine Disease Control Rate (PR+CR+Stable Disease (SD))
Evaluate PFS | 2 years
  Progression free survival in months
Evaluate Duration of Response, if any | 2 years
  Duration of Response (CR, PR, SD) in months

CONTACTS AND LOCATIONS:
Overall Officials: Steve Bernstein, MD, Study Director — Turnstone Biologics

IPD SHARING:
Plan to Share IPD: No